CLINICAL TRIAL: NCT05532787
Title: Comparison of Accelerated Diagnostic Pathways for Acute Chest Pain (EDACS & HEART Pathway) in Emergency Departments of the United Arab Emirates: A Multi-Center Prospective Study
Brief Title: Comparison of Accelerated Diagnostic Pathways for Acute Chest Pain in Emergency Departments in the United Arab Emirates
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zayed Military Hospital (Other Government)
Responsible Party: Principal Investigator, Farya Rehman, Emergency Medicine Post graduate year 4 Resident Doctor, Zayed Military Hospital
Other Study IDs: EDACS vs HEART pathway in UAE
Record Dates: First submitted 2022-09-03; First posted 2022-09-08 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Acute Coronary Syndrome; Chest Pain
MeSH Terms: conditions — Acute Coronary Syndrome; Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chest pain: Patients >18 years of age presenting to ED with chief complaint of chest pain or cardiac symptoms suggestive of acute coronary syndrome with at least one troponin ordered, without evidence of ST-segment elevation myocardial infarction on ECG
  Interventions: Other: Application of acute chest pain risk stratification scores (HEART and EDACS)

INTERVENTIONS:
Other: Application of acute chest pain risk stratification scores (HEART and EDACS) — Collection of data elements for the HEART Pathway and EDACS-ADP assessments and calculation of scores to risk stratify patients into low risk or high risk

SUMMARY:
This is a prospective four-site cohort study, which will accrue adults with symptoms concerning for acute coronary syndrome over a period of 12 months. After application of inclusion and exclusion criteria, Physicians will complete HEART Pathway and EDACS risk assessments on eligible participants. Major adverse cardiac events as defined by our study will be assessed at 30 days using electronic health record, telephone contact, and national death and health events search. Outcomes for all patients will then be matched against the existing pathway of care for acute chest pain that is being used currently to compare diagnostic accuracy of both scores to diagnose low risk chest pain in this population. The objective of this study is to compare the test performance of the HEART and EDACS pathway in a large cohort of patients presenting to the Emergency department with chest pain in the United Arab Emirates and to determine if either accelerated diagnostic pathway can achieve a negative predictive value of ≥99% for 30-day MACE as well as to externally validate EDACS-ADP and the HEART pathway in the UAE population and gain further insight into the applicability of these decision-making aids in different clinical settings in order to assess which score is best suitable for the UAE population. Our third objective is to compare the effectiveness of both scores to the existing framework for chest pain work up in each hospital and have the opportunity to unify Emergency Departments in their chest pain pathways in the UAE. The investigators will be testing the null hypothesis that there is no difference in using the EDACS-ADP to safely classify patients to low-risk category and early discharge from the ED versus the HEART pathway.

DETAILED DESCRIPTION:
The aim is to evaluate the safety, efficacy and economic feasibility of applying the EDACS and HEART pathways into existing EDs in the emirate of Abu Dhabi, UAE as well as to validate the sensitivity and NPV of these pathways given the United Arab Emirate's diverse population.

Over a period of 12 months, ED Physicians at four institutions will collect and retrieve data from their encounters with patients presenting with chest pain. Participants will be recruited from the EDs of four hospitals in the SEHA health network including Zayed Military Hospital, Tawam Hospital, Shaikh Shakhbout Medical City and Cleveland Clinic Abu Dhabi. Our study will include all eligible patients aged 18 years and above presenting acutely from the community to the ED with the chief complaint of chest pain or cardiac symptoms suggestive of ACS as defined by the American Heart Association with at least one troponin ordered, without evidence of ST-segment elevation myocardial infarction on ECG will be included. Chest pain will be defined as anterior chest pain, any discomfort located on the anterior thorax between the suprasternal notch and the xiphoid process, using the posterior axillary line as the border between the anterior and posterior thorax. In accordance with American Heart Association case definitions, other suggestive cardiac symptoms include the presence of epigastric, neck, jaw, or arm pain, discomfort or pressure without an apparent noncardiac source will also be included.

Patients that will be excluded are patients younger than 18 years or older than 90 years of age, patients with acute ST-segment elevation on the initial ECG in at least 2 contiguous leads, Hemodynamic instability (pulse rate persistently greater than 100 or less than 50 beats/min or systolic blood pressure persistently below 90 mm Hg), clear traumatic or radiologically evident of non-cardiac etiology, terminal non-cardiac illness, pregnancy or anticipated difficulty in communication or follow up such as any patient with no fixed address or telephone number in the UAE, previous enrollment and incapability or unwillingness for consent.

Data elements for the HEART Pathway and EDACS-ADP assessments will be entered prospectively by physicians into an Electronic Health Records (EHR)-based clinical decision support tool as well as alternatively a Data Collection Sheet will also be provided. EDACS-ADP and HEART pathways scores will be retrospectively calculated by research investigators not directly involved in patient care and will be logged in the Data collection sheet for each patient. After 30 days, patients will be reviewed for MACE defined as death, cardiac arrest, emergency revascularization procedure (coronary artery bypass grafting, stent placement, or other percutaneous coronary intervention), cardiogenic shock, ventricular arrhythmia needing intervention, high-degree atrioventricular block needing intervention, and acute myocardial infarction. All patients will undergo follow up by all three of the following approaches: telephone contact, review of patient hospital notes, and national death and health events search.

Data will be collected for a period of approximately 12 months from September onward, with a target sample size of 800 patients. Patients will be informed of the use of their de-identified data for research purposes and consented for its use. Informed written consent will be obtained from all subjects. All patient data will be anonymous and given a unique research ID. The data will be stored in an encrypted file on a secure computer, and all patient data will be protected. Extracted data from collection sheets will be stored on an encrypted hard drive, accessible only to investigators listed (as in the IRB form) and analyzed using the SPSS software.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 year old with a chief complaint of chest pain or cardiac symptoms (epigastric, neck, jaw, or arm pain, discomfort or pressure without an apparent noncardiac source).
* Greater than 18 year old chest pain/cardiac symptom patient with atleast one troponin ordered.

Exclusion Criteria:

* younger than 18 years
* older than 90 years of age
* acute ST-segment elevation on the initial ECG in at least 2 contiguous leads.
* Hemodynamic instability (pulse rate persistently greater than 100 or less than 50 beats/min or systolic blood pressure persistently below 90 mm Hg)
* clear traumatic or radiologically evident of non-cardiac etiology
* terminal non-cardiac illness
* pregnancy
* anticipated difficulty in communication or follow up
* previous enrollment
* incapability or unwillingness for consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients presenting with symptoms of chest pain or cardiac symptoms to the Emergency Department at Zayed Military Hospital, Tawam Hospital, Shaikh Shakhbout Medical City and Cleveland Clinic Abu Dhabi in the United Arab Emirates
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-02-03 (Actual); Primary Completion 2023-02-03 (Estimated); Study Completion 2023-03-03 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiac events | 30 days from initial patient encounter
  30 day major adverse cardiac event defined as death, cardiac arrest, emergency revascularization procedure (coronary artery bypass grafting, stent placement, or other percutaneous coronary intervention), cardiogenic shock, ventricular arrhythmia needing intervention, high-degree atrioventricular block needing intervention, and acute myocardial infarction.

CONTACTS AND LOCATIONS:
Overall Officials: Farya Rehman, MBBS, Principal Investigator — Zayed Military Hospital; Rauda Al Nuami, MBBS, Study Chair — Zayed Military Hospital
Locations (5):
- United Arab Emirates (5):
  - Cleveland Clinic Abu Dhabi, Abu Dhabi
  - Sheikh Khalifa Medical City, Abu Dhabi
  - Sheikh Shakhbout Medical City, Abu Dhabi
  - Zayed Military Hospital, Abu Dhabi
  - Tawam Hospital, Al Ain City

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers. Data will only be accessed and seen by the co-investigators listed in this research.

REFERENCES:
- [Background] Al-Shamsi S, Regmi D, Govender RD. Incidence of cardiovascular disease and its associated risk factors in at-risk men and women in the United Arab Emirates: a 9-year retrospective cohort study. BMC Cardiovasc Disord. 2019 Jun 17;19(1):148. doi: 10.1186/s12872-019-1131-2. PMID 31208354
- [Background] Eslick GD, Jones MP, Talley NJ. Non-cardiac chest pain: prevalence, risk factors, impact and consulting--a population-based study. Aliment Pharmacol Ther. 2003 May 1;17(9):1115-24. doi: 10.1046/j.1365-2036.2003.01557.x. PMID 12752348
- [Background] Litt HI, Gatsonis C, Snyder B, Singh H, Miller CD, Entrikin DW, Leaming JM, Gavin LJ, Pacella CB, Hollander JE. CT angiography for safe discharge of patients with possible acute coronary syndromes. N Engl J Med. 2012 Apr 12;366(15):1393-403. doi: 10.1056/NEJMoa1201163. Epub 2012 Mar 26. PMID 22449295
- [Background] Than M, Flaws D, Sanders S, Doust J, Glasziou P, Kline J, Aldous S, Troughton R, Reid C, Parsonage WA, Frampton C, Greenslade JH, Deely JM, Hess E, Sadiq AB, Singleton R, Shopland R, Vercoe L, Woolhouse-Williams M, Ardagh M, Bossuyt P, Bannister L, Cullen L. Development and validation of the Emergency Department Assessment of Chest pain Score and 2 h accelerated diagnostic protocol. Emerg Med Australas. 2014 Feb;26(1):34-44. doi: 10.1111/1742-6723.12164. Epub 2014 Jan 15. PMID 24428678
- [Background] Chapman AR, Lee KK, McAllister DA, Cullen L, Greenslade JH, Parsonage W, Worster A, Kavsak PA, Blankenberg S, Neumann J, Sorensen NA, Westermann D, Buijs MM, Verdel GJE, Pickering JW, Than MP, Twerenbold R, Badertscher P, Sabti Z, Mueller C, Anand A, Adamson P, Strachan FE, Ferry A, Sandeman D, Gray A, Body R, Keevil B, Carlton E, Greaves K, Korley FK, Metkus TS, Sandoval Y, Apple FS, Newby DE, Shah ASV, Mills NL. Association of High-Sensitivity Cardiac Troponin I Concentration With Cardiac Outcomes in Patients With Suspected Acute Coronary Syndrome. JAMA. 2017 Nov 21;318(19):1913-1924. doi: 10.1001/jama.2017.17488. PMID 29127948
- [Background] Chapman AR, Anand A, Boeddinghaus J, Ferry AV, Sandeman D, Adamson PD, Andrews J, Tan S, Cheng SF, D'Souza M, Orme K, Strachan FE, Nestelberger T, Twerenbold R, Badertscher P, Reichlin T, Gray A, Shah ASV, Mueller C, Newby DE, Mills NL. Comparison of the Efficacy and Safety of Early Rule-Out Pathways for Acute Myocardial Infarction. Circulation. 2017 Apr 25;135(17):1586-1596. doi: 10.1161/CIRCULATIONAHA.116.025021. Epub 2016 Dec 29. PMID 28034899
- [Background] Shin YS, Ahn S, Kim YJ, Ryoo SM, Sohn CH, Kim WY. External validation of the emergency department assessment of chest pain score accelerated diagnostic pathway (EDACS-ADP). Am J Emerg Med. 2020 Nov;38(11):2264-2270. doi: 10.1016/j.ajem.2019.09.019. Epub 2019 Nov 15. PMID 31757670
- [Background] Hess EP, Brison RJ, Perry JJ, Calder LA, Thiruganasambandamoorthy V, Agarwal D, Sadosty AT, Silvilotti ML, Jaffe AS, Montori VM, Wells GA, Stiell IG. Development of a clinical prediction rule for 30-day cardiac events in emergency department patients with chest pain and possible acute coronary syndrome. Ann Emerg Med. 2012 Feb;59(2):115-25.e1. doi: 10.1016/j.annemergmed.2011.07.026. Epub 2011 Sep 1. PMID 21885156
- [Background] Than MP, Pickering JW, Aldous SJ, Cullen L, Frampton CM, Peacock WF, Jaffe AS, Goodacre SW, Richards AM, Ardagh MW, Deely JM, Florkowski CM, George P, Hamilton GJ, Jardine DL, Troughton RW, van Wyk P, Young JM, Bannister L, Lord SJ. Effectiveness of EDACS Versus ADAPT Accelerated Diagnostic Pathways for Chest Pain: A Pragmatic Randomized Controlled Trial Embedded Within Practice. Ann Emerg Med. 2016 Jul;68(1):93-102.e1. doi: 10.1016/j.annemergmed.2016.01.001. PMID 26947800
- [Background] Stopyra J, Snavely AC, Hiestand B, Wells BJ, Lenoir KM, Herrington D, Hendley N, Ashburn NP, Miller CD, Mahler SA. Comparison of accelerated diagnostic pathways for acute chest pain risk stratification. Heart. 2020 Jul;106(13):977-984. doi: 10.1136/heartjnl-2019-316426. Epub 2020 Apr 8. PMID 32269131